CLINICAL TRIAL: NCT01042314
Title: A Study of the Effect of Concomitant Administration of BMS-708163 on the Pharmacokinetics of Donepezil in Healthy Subjects
Brief Title: Drug-Drug Interaction Study With Aricept® (Donepezil)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CN156-008
Record Dates: First submitted 2009-12-22; First posted 2010-01-05 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; BMS 708163

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Donepezil and BMS-708163 (Experimental)
  Interventions: Drug: Donepezil; Drug: BMS-708163

INTERVENTIONS:
Drug: Donepezil — Tablets, Oral, 5 mg, Once Daily, Days 1-28
  Other Names: Aricept®
Drug: BMS-708163 — Capsule, Oral, 125 mg, Once Daily, Days 15-28

SUMMARY:
The purpose of this study is to find out if the plasma concentration of donepezil is changed when BMS-708163 is administered at the same time

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and postmenopausal women

Exclusion Criteria:

* Medical History and Concurrent Diseases
* Gastrointestinal disease
* Gastrointestinal bleeding disorders
* History of peptic ulcer disease
* History of cholecystectomy
* History of seizure disorder
* History of asthma
* History of Chronic Obstructive Pulmonary Disease
* History of cardiac conduction abnormalities, including but not limited to "sick sinus syndrome" and those with unexplained syncopal episodes
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Aricept® alone and with BMS-708163: Aricept® Multiple-dose pharmacokinetic parameters (Cmax, Tmax, AUC (TAU), and Ctrough) will be assessed without BMS-708163 on Day 14 and with BMS-708163 (Ctrough) on Day 28 | Days 14 and 28

SECONDARY OUTCOMES:
Aricept® alone and with BMS-708163: Safety and tolerability based on adverse events, ECG, vital signs and safety labs | Days 7, 14, 21, 29 and study discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Parexel International - Baltimore Epcu, Baltimore, Maryland, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx